CLINICAL TRIAL: NCT00865670
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Geneva 600 mg Azithromycin Monohydrate Tablets and Pfizer Inc. (Zithromax) 600 mg Azithromycin Dihydrate Tablets in Healthy Adult Volunteers Under Fed Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Azithromycin 600 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA03414
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-03

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Azithromycin

ARMS (2):
- 1 (Experimental): Azithromycin Monohydrate 600mg Tablets
  Interventions: Drug: Azithromycin Monohydrate 600 mg Tablets
- 2 (Active Comparator): Zithromax (azithromycin dihydrate)600mg Tablets
  Interventions: Drug: Zithromax (azithromycin dihydrate) 600 mg Tablets

INTERVENTIONS:
Drug: Azithromycin Monohydrate 600 mg Tablets
  Arms: 1
Drug: Zithromax (azithromycin dihydrate) 600 mg Tablets
  Arms: 2

SUMMARY:
To demonstrate the bioequivalence of Azithromycin 600 mg Tablets Under Fed Conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C
* Treatment for drug or alcohol dependence
* Female subjects who are pregnant or lactating

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2003-08; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence according to US FDA guidelines | 32 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan S. Marion, M.D., Principal Investigator — MDS Pharma Services